CLINICAL TRIAL: NCT05462366
Title: Omics Sequencing of Specimen Derived From Mother-Infant-Pairs
Status: Recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Ma Ying, Clinical Professor, Zhujiang Hospital
Other Study IDs: ZhujiangHFCYXZX
Record Dates: First submitted 2022-07-06; First posted 2022-07-18 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Healthy; Breast-milk Collection; Feces
MeSH Terms: conditions — Breast Milk Expression | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Breastmilk and feces from mother-infant-pairs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mother: healthy mothers
  Interventions: Other: Sample collection
- Infant: healthy infants
  Interventions: Other: Sample collection

INTERVENTIONS:
Other: Sample collection — Collect breast-milk and feces from mother-infant-pairs.

SUMMARY:
The investigators aim to collect breast-milk and feces from the participants, and apply culture techniques as well as omics sequencing technology to probe into the microbial and metabolomic signature of the specimens.

ELIGIBILITY:
Inclusion Criteria:

* healthy pregnant women aged between 20y and 40y.
* Vaginal birth
* BMI<23.5 before pregnancy
* Infants' birth weight, between 2500g and 4000g.

Exclusion Criteria:

* gestational diabetes
* diagnosis of depressive disorder during pregnancy
* gestational hypertension
* diagnosis of other diseases during pregnancy
* Under probiotics or antibiotic treatment from 3 months prior to pregnancy till 3 months after delivery
* histrory of smoking and drinking alcohol
* history of diarrhea from 3 months prior to pregnancy till 3 months after delivery

Max Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This study intends to screen pregnant women in the Obstetrics and Gynecology Center of Zhujiang Hospital, Southern Medical University, and preliminarily recruit subjects that meet the inclusion criteria according to clinical diagnosis and auxiliary examination results. According to the specific conditions of vaginal delivery and post-birth newborns, the final inclusion of healthy pregnant women and newborns will be determined, and a total of 40-50 mother-infant-pairs will be recruited
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-22 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Compare the omics differences of the specimens between the experimental and control groups | 2021.7.1-2026.12.30
  Apply 16S amplicon sequencing and shotgun sequencing technology to obtain microbial structure of the specimens. The differences of microbial structure will be compared between the experimental and control groups. Significance among multiple groups was tested using a one-way analysis of variance (ANOVA), followed by the least significant difference (LSD) post hoc test. Groups with different characters denoting a significant difference, while having the same character denotes p-value > 0.05 in LSD test.
Compare the microbial feature differences of the specimens between the experimental and control groups | 2021.7.1-2026.12.30
  Apply traditional culture technologies to validate and obtain human source bacteria.The differences of frequencies of probiotics will be compared between the experimental and control groups. Depending on the distribution of the variables, either the Mann-Whitney test or the unpaired Student's t-test was employed for quantitative variables. The Kruskal-Wallis test for mean values was used to evaluate non-parametric comparisons between participants in all groups. Significance among multiple groups was tested using a one-way analysis of variance (ANOVA), followed by the least significant difference (LSD) post hoc test. Groups with different characters denoting a significant difference, while having the same character denotes p-value > 0.05 in LSD test.

SECONDARY OUTCOMES:
Compare the health status differences between the experimental and control groups | 2021.7.1-2026.12.30
  After a brief introduction to the survey, participants were asked to complete a questionnaire. The differences of health status will be compared between the experimental and control groups. Depending on the distribution of the variables, either the Mann-Whitney test or the unpaired Student's t-test was employed for quantitative variables. The Kruskal-Wallis test for mean values was used to evaluate non-parametric comparisons between participants in all groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided